CLINICAL TRIAL: NCT03298360
Title: A Chronological Study of the Formation of HIV Cellular Reservoirs Through the Expression of Surface Markers on CD4 + T Lymphocytes, Including CD32a
Acronym: ANRS EP63
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS EP63 RESTA 32a
Record Dates: First submitted 2017-09-20; First posted 2017-10-02 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: HIV Infections
Keywords: HIV cell reservoir
MeSH Terms: conditions — HIV Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood sample — 167mL of blood in EDTA tube will be obtained on a research visit, after signature of written informed consent

SUMMARY:
To analyze the HIV viral sequences present in the CD32 + CD4a + T lymphocytes of the patients who have participated in the ANRS 139 TRIO trial, always followed and in virological success, and carrying multi-resistant viruses archived in the HIV cell reservoir, in order to reconstruct the chronology of the installation of this reservoir.

DETAILED DESCRIPTION:
Objectives

Principal objective

To analyze the HIV viral sequences present in the CD32 + CD4a + T lymphocytes of the patients who have participated in the ANRS 139 TRIO trial, always followed and in virological success, and carrying multi-resistant viruses archived in the HIV cell reservoir, in order to reconstruct the chronology of the installation of this reservoir.

Secondary objectives

To analyze the HIV viral sequences present in the CD4 + lymphocytes with other membrane HIV reservoir markers, currently being identified, in these same patients

Methodology

Pathophysiological study, in patients infected by multi drug-resistant viruses

Estimated enrollment

21 participants (total and per group)

Intervention

167mL blood sample in EDTA tube:

* 160mL (16 tubes of 10mL): for IGH (Institute of Human Genetics-Montpellier)
* 7mL (1tube of 7mL): to measure HIV-RNA in centers

Estimated planning or Study / Trial timetable

Study start date: September 2017

Enrollment period: 12 months

Total study duration: 24 months (analyses included)

Estimated study/trial completion date: September 2019 (one year after enrollment of the last patient)

Study design

Cross-sectional survey, 167mL of blood in EDTA tube will be obtained on a research visit, after signature of written informed consent

ELIGIBILITY:
Inclusion Criteria:

* Patients who participated to ANRS139 TRIO trial, and still followed in centers
* Who remained in virological success since the participation at the trial: 90% of HIV-1 RNA level less than 50 copies/mL : one or more blips less than 1000 copies/mL are tolerated
* Genotypic resistance profiles available at baseline and before trial
* Age ≥ 18 years
* Affiliate or beneficiary of a social security system (the State Medical Aid or AME is not a social security system).
* Written informed consent signed by the person and the investigator before any exam performed in the study.

Exclusion Criteria:

* HIV-1 RNA level ≥ 1000 copies/mL at least once since the end of the 139 TRIO trial
* Patient participating in another research evaluating other treatments with an exclusion period ongoing at the screening visit.
* Person under legal guardianship or deprived of liberty by a judicial or administrative decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV Infection
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Presence of HIV viral sequences in the CD32 + CD4a + T lymphocytes of the patients | inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Monsef BENKIRANE, Montpellier, France